CLINICAL TRIAL: NCT02404779
Title: Treatment of Intracranial Hypertension of Severe Tramatic Brain Injured Patients. Physiopathologic Effects of Neuromuscular Blocking Agents. A Controlled Randomized Study Versus Placebo
Brief Title: Treatment of Intracranial Hypertension of Severe Tramatic Brain Injured Patients. Physiopathologic Effects of Neuromuscular Blocking Agents
Acronym: THIC Cu
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0225; 2014-004951-30 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-04-01 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
Keywords: ICU; Deep sedation; Mechanical ventilation; Traumatic brain injury; Intracranial hypertension; Cisatracurium; Neuromuscular Blocking Agent; Randomization versus placebo
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — cisatracurium

ARMS (2):
- CISATRACURIUM (Experimental): To compare the evolution of intracranial pressure (ICP) of severely brain injured patients with intracranial hypertension after administration of cisatracurium versus placebo.
  Interventions: Drug: cisatracurium besilate
- PLACEBO (Placebo Comparator): To compare the evolution of intracranial pressure (ICP) of severely brain injured patients with intracranial hypertension after administration of cisatracurium versus placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: cisatracurium besilate
  Arms: CISATRACURIUM
Other: Placebo
  Arms: PLACEBO

SUMMARY:
Severely brain injured patients are at high risk of intracranial hypertension. Among medical treatments (sedatives), neuromuscular blocking agents (NMBA) are recommended by french but not english speaking societies.

Effects of NMBA are unknown. The present study is designed to compare the effects of NMBA versus placebo in the treatment of intracranial hypertension, and the underlying physiopathologic effects.

DETAILED DESCRIPTION:
In case of intracranial hypertension, french neurocritical care society argue for the use of neuromuscular blocking agents before osmotherapy, barbituric coma, hypothermia and craniectomy.

English speaking societies don't sustain this approach. Since then, the use of NMBA remains controversial in case of intracranial hypertension and no study is available.

We propose to study severely brain injured patients presenting with intracranial hypertension and treat them with cisatracurium besilate or placebo.

Our hypothesis is that neuromuscular blockade might act on several parameters:

* Hemodynamics
* respiratory parameters, mechanical ventilation and blood gaz analysis
* cerebral velocities
* diminished O2 peripheral consumption
* cerebrospinal diffusion and concentration of cisatracurium and a metabolite laudanosine We wish to assess changes in ICP according to the above parameters in a controlled randomized non blinded fashion against placebo (NaCl 0,9%).

ELIGIBILITY:
Inclusion Criteria:

* - Age over 18
* Mechanical ventilation and deep sedation
* Severe traumatic brain injury
* Intracranial hypertension (ICP > 20 mmHg during > 15 minutes)
* Intracranial pressure monitoring
* Hemodynamically stable

Exclusion Criteria:

* - History of anaphylaxia with neuromuscular agents
* Hemodynamic instability
* Pregnant and/or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-03-19 (Actual); Primary Completion 2022-03-19 (Estimated); Study Completion 2022-06-18 (Estimated)

PRIMARY OUTCOMES:
area under the curve of the temporal evolution of intracranial pressure | at day 1
  The primary outcome is the area under the curve of the temporal evolution of intracranial pressure, over a period of 30 minutes after the administration of neuromuscular blocking agent or placebo.

SECONDARY OUTCOMES:
Course of intracranial and cerebral perfusion pressures and various cerebral monitoring data if available (SvjO2, PtiO2) | at day 1
Monitoring of the time spent by intracranial pressure above 20 mmHg using continuous recording | at day 1
Course of intracranial pressure based on the type of brain injury | at day 1
  diffuse axonal injury, subarachnoid hemorrhage, intracerebral hematoma)
Monitoring of the curare effect | at day 1
  train of four and PTC
Course of ventilation parameters | at day 1
  tidal volume, FiO2, PEEP
Course of transcranial Doppler data | at day 1
  velocities
Course of arterial blood gas data | at day 1
  pH, paO2, paCO2, Excess Base, HCO3-
Course of plasma and cerebrospinal fluid concentrations of cistracurium and laudanosine | at day 1
Cerebrospinal fluid concentrations of cisatracurium and laudanosin in case of cerebrospinal fluid derivation | at day 1
Occurrence of cardiovascular complications | at day 1
  hypotension, myocardial ischemia
Occurrence of pulmonary complications | at day 1
  acute respiratory distress syndrome, pneumonia acquired under mechanical ventilation
Occurrence of renal complications | at day 1
  use of renal replacement therapy
Occurrence of infectious complications | at day 1
Doses of vasopressors or catecholamines | at day 1
Need to increase therapeutics | at day 1
  barbiturate coma, hypothermia, osmotherapy, decompressive craniectomy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France